CLINICAL TRIAL: NCT02265796
Title: Improvement of Subjective Well-Being by Ranolazine Among Unrevascularized Chronic Stable Coronary Artery Disease Patients
Brief Title: Ranolazine Among Unrevascularized Chronic Stable Angina Patients
Acronym: IMWELL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: North Florida Foundation for Research and Education (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Anthony A Bavry, Interventional Cardiologist, North Florida Foundation for Research and Education
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 149-2013
Record Dates: First submitted 2014-10-10; First posted 2014-10-16 (Estimated); Results first posted 2017-12-04 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Angina
Keywords: deferred percutaneous coronary intervention; fractional flow reserve
MeSH Terms: conditions — Angina Pectoris | interventions — Ranolazine; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ranolazine (Active Comparator): Ranolazine 500 mg tablets
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Interventions: Drug: Ranolazine
- Sugar pill (Placebo Comparator): Sugar pill that looks like the drug ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Ranolazine — Ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Other Names: Ranexa
  Arms: Ranolazine
Drug: Sugar pill — 1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Other Names: placebo
  Arms: Sugar pill

SUMMARY:
This is a prospective, double-blind, placebo-controlled, randomized, single-center (North Florida- South Georgia VA Medical Center) study. The study objective is to determine if ranolazine improves angina symptoms at 4 months compared with placebo among stable coronary artery disease patients who have demonstrable myocardial ischemia, but who do not undergo revascularization

DETAILED DESCRIPTION:
This is a prospective, double-blind, placebo-controlled, randomized, single-center (North Florida- South Georgia VA Medical Center) study. The study objective is to determine if ranolazine improves angina symptoms at 4 months compared with placebo among stable coronary artery disease patients who have demonstrable myocardial ischemia, but who do not undergo revascularization.

Baseline Procedure:

Assessments performed exclusively to determine eligibility for this study would be done only after obtaining informed consent. Assessments performed for clinical indications (not exclusively to determine study eligibility) may be used for baseline values even if the studies were done before informed consent was obtained. The assessment will include:

* Informed Consent
* Review subject eligibility criteria
* FFR value calculated at the time of cardiac catheterization
* Review previous and concomitant medications
* Frequency of symptoms and quality of life prior to study according to Seattle Angina Questionnaire (SAQ)

Screening Visit:

The assessments to determine eligibility are:

* Review of eligibility criteria
* Review of cardiac catheterization and FFR
* Review of medications taken in the past 30 days Subjects that meet eligibility criteria will be randomized to receive either the active drug, Ranolazine or a matching placebo (non-active drug). Staff and subjects will not know if the subject will be receiving the active drug or the placebo.

Drug schedule will be as follows:

* 1st dose of one tablet (500mg) will begin the evening of Day 1
* On Days 2-7, one tablet (500mg) two times a day (12-hours apart).
* On Day 8, increase dose of study drug to two tablets (1000mg) twice a day; once in the morning and once in the evening, 12 hours apart. This dose will continue for the duration of the study. The study drug can be taken with or without food.

Telephone Follow-up:

One week phone calls will be made to determine well being, adverse events, answer questions and remind subjects to increase the study medication dose.

Month 4 Follow-up:

* Frequency of symptoms and quality of life according to Seattle Angina Questionnaire (SAQ)
* Assessment of well-being
* Any hospitalizations or the need for revascularization

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >= 18 years of age referred for cardiac catheterization for evaluation of cardiac symptoms ( angina, fatigue, or shortness of breath)
* At least 1 indeterminate stenosis (20-80%),
* Fractional flow reserve (FFR) <=0.8 and PCI deferred

Exclusion Criteria:

* Coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) during the index procedure or anticipated within the next month
* acute coronary syndrome or cardiogenic shock
* QTc > 500 milliseconds
* use of strong inhibitors of CTP3A (i.e. ketoconazole, itraconazole, clarithromycin,nefazodone, nelfinavir, ritonavir, indinavir and saquinavir)
* use of inducers of CYP3A (i.e. rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine, and St. John's wort)
* liver cirrhosis
* sever renal insufficiency (i.e. creatinine clearance < 30mL/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Bavry, MD, MPH, Principal Investigator — NorthFlorida/South Georgia Veterans Health System, Gainesville, FL 32608
Locations (1):
- North Florida/South Georgia Veterans Health System, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bavry AA, Park KE, Choi CY, Mahmoud AN, Wen X, Elgendy IY. Improvement of Subjective Well-Being by Ranolazine in Patients with Chronic Angina and Known Myocardial Ischemia (IMWELL Study). Cardiol Ther. 2017 Jun;6(1):81-88. doi: 10.1007/s40119-016-0081-3. Epub 2017 Jan 2. PMID 28044265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period first subject enrolled 9/24/2014 to last subject enrolled 12/12/2015
Groups:
- Ranolazine: Ranolazine 500 mg tablets
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Ranolazine: Ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
- Sugar Pill: Sugar pill that looks like the drug ranolazine 500mg tablet
  1. 500mg tablet two times per day for 7 days then,
  2. 500mg tablet (1000mg) two times per day for 15 weeks
  Sugar pill: 1. 500mg tablet two times per day for 7 days then, 2. 500mg tablet (1000mg) two times per day for 15 weeks
Period: Overall Study
Arm/Group | Ranolazine | Sugar Pill
Started | 25 | 25
Completed | 22 | 24
Not Completed | 3 | 1
Not completed — Death | 1 | 0
Not completed — started on excluded medication | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Sugar Pill | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 15 | 13 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 24 | 25 | 49
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50
Hypertension [Count of Participants; unit: Participants] | 25 | 25 | 50
Hyperlipidemia [Count of Participants; unit: Participants] | 16 | 17 | 33
Diabetes mellitus [Count of Participants; unit: Participants] | 14 | 16 | 30
on Insulin [Count of Participants; unit: Participants] | 5 | 7 | 12
history of Percutaneous Coronary Intervention [Count of Participants; unit: Participants] | 19 | 14 | 33
history of Coronary Artery Bypass Graft surgery [Count of Participants; unit: Participants] | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Seattle Angina Questionnaire Score Change From Baseline to 16 Weeks
Description: The SAQ quantifies patients' physical limitations caused by angina, the frequency of and recent changes in their symptoms, their satisfaction with treatment, and the degree to which they perceive their disease to affect their quality of life.Each of the 5 dimensions are scored by assigning eachresponse an ordinal value, beginning with 1 for the response that implies the lowest level of functioning, and summing across items within each of the 5 scales. Scale scores then transformed to 0-100 range by subtracting the lowest possible scale score, dividing by the range1 / 3 Seattle Angina Questionnaire (SAQ)of the scale and multiplying by 100. No overall scale score is generated.
  Factors and Each scale is transformed to a score of 0 to 100, where higher scores indicate better function (eg, less physical limitation, less angina, and better quality of life).
  .
Time Frame: Change in baseline to 16 weeks
Population: by intention to treat, 46 subjects had baseline and follow up SAQ data completed at 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranolazine | Sugar Pill
Number analyzed (Participants) | 22 | 24
units on a scale
  Physical Limitation baseline | 48 (25) | 50 (20)
  Physical Limitation 16 weeks | 40 (19) | 60 (24)
  Physical Limitation group difference | -7 (27) | 6 (20)
  Angina Stability baseline | 39 (28) | 37 (28)
  Angina Stablility 16 weeks | 58 (26) | 55 (27)
  Angia Stability group difference | 19 (36) | 18 (32)
  Angina Frequency baseline | 65 (24) | 64 (23)
  Angina Frequency 16 weeks | 81 (23) | 80 (24)
  Angina Frequency group difference | 16 (36) | 15 (27)
  Treatment Satisfaction baseline | 80 (19) | 85 (18)
  Treatment Statisfaction 16 weeks | 77 (26) | 82 (22)
  Treatment Satisfaciton group difference | -4 (26) | -3 (26)
  Quality of Life baseline | 37 (24) | 45 (27)
  Quality of Life 16 weeks | 56 (29) | 63 (18)
  Quality of Life group difference | 21 (32) | 18 (31)
Statistical Analysis 1: Comparison: Ranolazine vs Sugar Pill; between group comparison for all SAQ domains; Test type: Superiority; p > 0.05, t-test, 2 sided — the reported p value is for all between group comparisons of the SAQ domains
Statistical Analysis 2: Comparison: Ranolazine; within group comparison of change from baseline; Test type: Superiority; p > 0.05, paired t test — reported p value is for the physical limitation, angina frequency and treatment satisfaction domains
Statistical Analysis 3: Comparison: Ranolazine; within group comparison of change from baseline; Test type: Superiority; p < 0.05, paired t test — reported p value is for the angina stability and quality of life domains
Statistical Analysis 4: Comparison: Sugar Pill; within group comparison of change from baseline; Test type: Superiority; p > 0.05, paired t test — reported p value is for the physical limitation and treatment satisfaction domains
Statistical Analysis 5: Comparison: Sugar Pill; within group comparison of change from baseline; Test type: Superiority; p < 0.05, paired t test — reported p value is for the angina stability, angina frequency and quality of life domains

2. Secondary Outcome: Subjective Well Being
Description: overall feeling of well being determined from rating of excellent, good, fair or poor at baseline compared to same at month 4
Time Frame: Compare from baseline to month 4
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Sugar Pill
Number analyzed (Participants) | 22 | 24
Participants
  Baseline: excellent/good | 9 | 6
  Baseline: fair/poor | 12 | 16
  Baseline: missing | 1 | 2
  16 Weeks: excellent/good | 11 | 10
  16 Weeks: fair/poor | 10 | 10
  16 Weeks: missing | 1 | 4
Statistical Analysis 1: Comparison: Ranolazine vs Sugar Pill; between group comparison for the "excellent/good"; Test type: Superiority; p = 0.58, Fisher Exact
Statistical Analysis 2: Comparison: Ranolazine vs Sugar Pill; Between group analysis for "fair/poor"; Test type: Superiority; p = 0.80, Fisher Exact
Statistical Analysis 3: Comparison: Ranolazine; within group analysis of change from baseline for excellent/good; Test type: Superiority; p = 0.50, McNemar
Statistical Analysis 4: Comparison: Ranolazine; within group comparison of change from baseline for fair/poor; Test type: Superiority; p = 0.48, McNemar
Statistical Analysis 5: Comparison: Sugar Pill; within group analysis of change from baseline for excellent/good; Test type: Superiority; p = 0.19, McNemar
Statistical Analysis 6: Comparison: Sugar Pill; within group comparison of change from baseline for fair/poor; Test type: Superiority; p = 0.067, McNemar

3. Secondary Outcome: Ischemia Driven Revascularization or Hospitalization
Description: Number of participants who reported adverse events for ischemia driven revascularization or hospitalization
Time Frame: 4 month
Population: the incidence of ischemia driven hospitalization or catheterization was assessed for all subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Sugar Pill
Number analyzed (Participants) | 25 | 25
Participants | 3 | 5
Statistical Analysis 1: Comparison: Ranolazine vs Sugar Pill; Test type: Superiority; p > 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline to 16 weeks
Description: adverse events assessed at 1 week, 4 week and 16 week phone call follow-up.
Arm/Group | Ranolazine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 5/25 | 4/25
Other Adverse Events (participants affected / at risk) | 17/25 | 15/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=25) | Sugar Pill (N=25)
lung mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
death (Cardiac disorders) | 1 (1) | 0 (0)
bradycardia, symptomatic (Cardiac disorders) | 1 (1) | 0 (0)
Unstable Angina (Cardiac disorders) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Myocardial Infarctoin (Cardiac disorders) | 1 (1) | 0 (0)
chest pain (Cardiac disorders) | 1 (1) | 0 (0)
coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) — Coronary artery bypass surgery
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=25) | Sugar Pill (N=25)
anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
dizziness (Nervous system disorders) | 5 (5) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fainting (Nervous system disorders) | 3 (3) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
worsening renal function (Renal and urinary disorders) | 1 (1) | 0 (0)
Leg cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Black stools (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No